CLINICAL TRIAL: NCT00333476
Title: A Phase 2, Randomized, Open Label, Safety, and Pharmacodynamic Study of Squalamine Lactate for Injection for the Treatment of Minimally Classic or Active Occult Choroidal Neovascularization Associated With Age-Related Macular Degeneration
Brief Title: A Study of MSI-1256F (Squalamine Lactate) To Treat "Wet" Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MSI-1256F-212
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — squalamine lactate

INTERVENTIONS:
Drug: MSI-1256F (Squalamine Lactate)

SUMMARY:
Age-Related Macular Degeneration (AMD) is a degenerative eye disease of the retina that causes a progressive loss of central vision. AMD is the leading cause of legal blindness among adults age 50 or older in the Western world. AMD presents in two different types - "dry" and the more severe "wet" form. Wet AMD is caused by the growth of abnormal blood vessels in the macula. Squalamine lactate is an investigational drug that may prevent the growth of these abnormal blood vessels. This study will test the safety and efficacy of Squalamine in the treatment of AMD.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 50 years of age.
* minimally classic or active occult choroidal neovascularization associated with age-related macular degeneration in one or both eyes.
* baseline best corrected visual acuity score between 35 to 65 letters according to the Early Treatment of Diabetic Retinopathy Study protocol.
* central retinal thickness by optical coherence tomography of > 250 microns.
* lesions > 9 disc areas.
* > 25% fibrosis in the lesion.

Exclusion Criteria:

* Previous history of triamcinolone, bevacizumab, ranibizumab, or pegaptanib sodium injection therapy in the study eye.
* retinal or optic nerve disease.
* uncontrolled diabetes.
* ongoing malignancy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2006-05

PRIMARY OUTCOMES:
To evaluate the safety profile of squalamine lactate at doses ranging from 40 mg to 160 mg of squalamine lactate

SECONDARY OUTCOMES:
To evaluate short-term effects on best corrected visual acuity and changes in subretinal CNV as measured by optical coherence tomography
To evaluate short-term effects on best corrected visual acuity and changes in subretinal CNV as measured by fluorescein angiography

CONTACTS AND LOCATIONS:
Overall Officials: Randy Katz, MD, Principal Investigator — Florida Eye Microsurgical Institute, Inc.; Alexander Eaton, MD, Principal Investigator — Retina Health Center; Thomas Ciulla, MD, Principal Investigator — Midwest Eye Institute; Raymond Sjaarda, MD, Principal Investigator — Retina Specialists; Nelson Sabates, MD, Principal Investigator — Eye Foundation of Kansas City; Charles Garcia, MD, Principal Investigator — Charles Garcia, MD, P.A.; Glenn Stoller, MD, Principal Investigator — Ophthalmic Consultants of Long Island; Phillip Rosenfeld, MD, Principal Investigator — Bascom Palmer Eye Institute; Steven Rose, MD, Principal Investigator — Retina Associates of Western New York
Locations (9):
- United States (9):
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Retina Health Center, Fort Meyers, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina Specialists, Towson, Maryland
  - Eye Foundation of Kansas City, Kansas City, Missouri
  - Ophthalmic Consultants of Long Island, Long Island City, New York
  - Retina Associates of Western New York, Rochester, New York
  - Charles Garcia, MD, P.A., Houston, Texas